CLINICAL TRIAL: NCT00772213
Title: The Impact of a Multifunctional Image Guided Therapy Suite (MIGTS) on Emergency Multiple Trauma Care - a Controlled Clinical Pilot Study
Brief Title: The Multifunctional Image Guided Therapy Suite (MIGTS) in Emergency Multiple Trauma Care
Acronym: MIGTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); Scientific Foundation of the Swiss Accident Insurance Fond (Unknown); Voluntary Academic Society, Basel (Unknown); CARCAS Switzerland (Unknown)
Responsible Party: Principal Investigator, Thomas Gross, Prof. Dr. med., University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK 159/02
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Acceleration of Procedure; Reduction of Number of Transports and Transfers; Involved Staff Member's Evaluation
Keywords: multiple trauma; outcome and process assessment
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MIGTS treatment (Experimental): controlled trial (quasi-randomized) versus controls (=conventional treatment not in the MIGTS)
  Interventions: Procedure: MIGTS treatment
- controls (=conventional treatment not in the MIGTS) (No Intervention)

INTERVENTIONS:
Procedure: MIGTS treatment — treatment of multiple trauma patients in the MIGTS
  Other Names: combined diagnostic and operation room
  Arms: MIGTS treatment

SUMMARY:
Controlled clinical intervention study comparing the treatment of multiple trauma patients in a newly developed combined diagnostic and operation room, the multifunctional image guided therapy suite (MIGTS) versus controls. The MIGTS proved to significantly accelerate the procedure and led to more satisfied team members.

DETAILED DESCRIPTION:
Objective: Pilot evaluation to which extend the implementation of a newly developed combined diagnostic and operation room, the multifunctional image guided therapy suite (MIGTS) may influence the emergency treatment of multiply injured patients.

Summary Background: Controlled data on the impact of modern technology integration in multiple trauma management and involved care providers are lacking.

Methods: Quasi-randomized clinical intervention study comparing the treatment of multiple trauma patients (injury severity score, ISS >16) in the MIGTS versus controls.

ELIGIBILITY:
Inclusion Criteria:

* multiple trauma with
* at least two abbreviated injury scoring (AIS) regions involved and
* injury severity score (ISS)>16
* primary hospital treatment at University Hospital Basel

Exclusion Criteria:

* monotrauma or
* ISS < 16 or
* prior treatment in another hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2003-02; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Time to first CT scan | first CT scan after arrival of emergency patient

SECONDARY OUTCOMES:
Staff member evaluation (Likert scale 1-5) | end of emergency treatment (arrival ICU or death)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gross, Prof. Dr., Principal Investigator — University of Basel
Locations (1):
- University Hospital, CARCAS group, Basel, Switzerland

REFERENCES:
- [Background] Messmer P, Jacob AL, Fries E, Gross T, Suhm N, Steinbrich W, Frede KE, Schneider T, Regazzoni P. [Technology integration and process management. Concept and implementation of a new platform for simultaneous diagnosis and therapy of acutely ill and injured patients and for elective computer assisted surgery (CAS)]. Unfallchirurg. 2001 Oct;104(10):1025-30. doi: 10.1007/s001130170047. German. PMID 11699300
- [Background] Gross T, Amsler F, Ummenhofer W, Zuercher M, Regazzoni P, Jacob AL, Huegli RW, Messmer P. [Interdisciplinary emergency room management of trauma patients from the standpoint of coworkers]. Chirurg. 2005 Oct;76(10):959-66. doi: 10.1007/s00104-005-1068-0. German. PMID 16021393
- [Result] Gross T, Messmer P, Amsler F, Fuglistaler-Montali I, Zurcher M, Hugli RW, Regazzoni P, Jacob AL. Impact of a multifunctional image-guided therapy suite on emergency multiple trauma care. Br J Surg. 2010 Jan;97(1):118-27. doi: 10.1002/bjs.6842. PMID 19937992
- See also: Related Info — http://carcas.wordpress.com